CLINICAL TRIAL: NCT00934609
Title: Effects of 12-weeks Endurance Training in Patients With Chronic Heart Failure Due to Dilated Cardiomyopathy
Brief Title: Training Study to Evaluate the Benefit of Exercise for Patients With Chronic Heart Failure
Acronym: CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Collaborators: The German Heart Foundation (Other)
Responsible Party: Prof. Dr. Tim Meyer, Institute of Sports- and Preventive Medicine, Saarland University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000-01SaarlandU
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Dilated Cardiomyopathy; Chronic Heart Failure
Keywords: Exercise; heart failure; dilated cardiomyopathy; Endurance training
MeSH Terms: conditions — Cardiomyopathy, Dilated; Motor Activity; Heart Failure | interventions — Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Experimental): 12 weeks of endurance training on the cycle ergometer under supervision on a physician
  Interventions: Behavioral: Endurance training
- Control (No Intervention): Control condition

INTERVENTIONS:
Behavioral: Endurance training — 45 min ergometer cycling at the ventilatory anaerobic threshold 4 times per week for 12 weeks
  Arms: Training

SUMMARY:
The study investigates the safety and effectiveness of a 12 week endurance training program for patients with chronic heart failure

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure NYHA stage 2 and 3

Exclusion Criteria:

* Valvular disease
* recent decompensation
* Other complaints that might interfere with ergometer exercise

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)

PRIMARY OUTCOMES:
Physical capacity

SECONDARY OUTCOMES:
Left ventricular function
occurence of complications | within study period

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports- and Preventive Medicine, Saarland University, Saarbrücken, Saarland, Germany